CLINICAL TRIAL: NCT01392326
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Study of Secukinumab to Demonstrate the Efficacy at 24 Weeks and to Assess the Long Term Safety, Tolerability and Efficacy up to 2 Years in Patients With Active Psoriatic Arthritis
Brief Title: Efficacy at 24 Weeks and Long Term Safety, Tolerability and Efficacy up to 2 Years of Secukinumab (AIN457) in Patients With Active Psoriatic Arthritis (PsA)
Acronym: FUTURE 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457F2306; 2011-000276-34 (EudraCT Number)
Record Dates: First submitted 2011-07-07; First posted 2011-07-12 (Estimated); Results first posted 2016-02-04 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-01

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic arthritis; PsA; ACR; CASPAR
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Experimental): Secukinumab (75mg)
  Interventions: Drug: Secukinumab (75 mg)
- Group 2 (Experimental): Secukinumab (150 mg)
  Interventions: Drug: Secukinumab (150 mg)
- Group 3 (Placebo Comparator)
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Secukinumab (75 mg) — Secukinumab (75 mg)
  Arms: Group 1
Drug: Secukinumab (150 mg) — Secukinumab (150 mg)
  Arms: Group 2
Drug: Placebo Comparator — Placebo Comparator
  Arms: Group 3

SUMMARY:
This study will assess the efficacy and safety of secukinumab in patients with active psoriatic arthritis who are intolerant to or have had an inadequate response to NSAIDs, DMARDs and / or TNFα inhibitor therapy.

ELIGIBILITY:
Inclusion criteria:

* Male or non-pregnant, non-lactating female patients at least 18 years of age
* Diagnosis of PsA classified by CASPAR criteria and with symptoms for at least 6 months with moderate to severe PsA who must have at Baseline ≥3 tender joints out of 78 and ≥3 swollen out of 76 (dactylitis of a digit counts as one joint each)
* Rheumatoid factor and anti-CCP antibodies negative
* Diagnosis of active plaque psoriasis, with at least one psoriatic plaque of ≥2cm diameter or nail changes consistent with psoriasis or documented history o plaque psoriasis

Exclusion criteria:

* Chest X-ray with evidence of ongoing infectious or malignant process
* Subjects who have previously been treated with more than 3 different TNFα inhibitors
* Subjects taking high potency opioid analgesics
* Subjects who have ever received biologic immunomodulating agents except for those targeting TNFα Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 606 (Actual)
Dates: Start 2011-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (94):
- United States (23):
  - Novartis Investigative Site, Anniston, Alabama
  - Novartis Investigative Site, Mesa, Arizona
  - Novartis Investigative Site, Paradise Valley, Arizona
  - Novartis Investigative Site, Upland, California
  - Novartis Investigative Site, Tamarac, Florida
  - Novartis Investigative Site, Newnan, Georgia
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Eagan, Minnesota
  - Novartis Investigative Site, Richmond Heights, Missouri
  - Novartis Investigative Site, Lincoln, Nebraska
  - Novartis Investigative Site, Freehold, New Jersey
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Duncansville, Pennsylvania
  - Novartis Investigative Site, Johnston, Rhode Island
  - Novartis Investigative Site, Columbia, South Carolina
  - Novartis Investigative Site, North Charleston, South Carolina
  - Novartis Investigative Site, Jackson, Tennessee
  - Novartis Investigative Site, Benbrook, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Mesquite, Texas
  - Novartis Investigative Site, Seattle, Washington
- Argentina (4):
  - Novartis Investigative Site, Buenos Aires, Buenos Aires
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, Córdoba, Córdoba Province
  - Novartis Investigative Site, Rosario, Santa Fe Province
- Australia (2):
  - Novartis Investigative Site, Maroochydore, Queensland
  - Novartis Investigative Site, Malvern, Victoria
- Belgium (3):
  - Novartis Investigative Site, Genk
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Leuven
- Brazil (2):
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, São Paulo, São Paulo
- Bulgaria (3):
  - Novartis Investigative Site, Sevlievo, Bulgaria
  - Novartis Investigative Site, Sofia, Bulgaria
  - Novartis Investigative Site, Pleven
- Canada (4):
  - Novartis Investigative Site, St. John's, Newfoundland and Labrador
  - Novartis Investigative Site, Newmarket, Ontario
  - Novartis Investigative Site, Waterloo, Ontario
  - Novartis Investigative Site, Trois-Rivières, Quebec
- Czechia (3):
  - Novartis Investigative Site, Bruntál, Czech Republic
  - Novartis Investigative Site, Uherské Hradiště, Czech Republic
  - Novartis Investigative Site, Zlín, Czech Republic
- Germany (12):
  - Novartis Investigative Site, Berlin, Germany
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Gommern
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Herne
  - Novartis Investigative Site, Hildesheim
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Ratingen
  - Novartis Investigative Site, Zerbst
- Israel (4):
  - Novartis Investigative Site, Ashkelon
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Italy (4):
  - Novartis Investigative Site, Valeggio sul Mincio, (vr)
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Prato, PO
  - Novartis Investigative Site, Siena, SI
- Philippines (7):
  - Novartis Investigative Site, Lipa City, Batangas
  - Novartis Investigative Site, Dasmariñas, Cavite
  - Novartis Investigative Site, Manila, National Capital Region
  - Novartis Investigative Site, Manila, Philippines
  - Novartis Investigative Site, Las Piñas
  - Novartis Investigative Site, Manila
  - Novartis Investigative Site, Quezon City
- Poland (2):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Warsaw
- Romania (4):
  - Novartis Investigative Site, Bucharest, District 1
  - Novartis Investigative Site, Iași, Iaşi
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Cluj-Napoca
- Russia (5):
  - Novartis Investigative Site, Kemerovo
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Yaroslavl
  - Novartis Investigative Site, Yekaterinburg
- Novartis Investigative Site, Singapore, Singapore, Singapore
- Slovakia (2):
  - Novartis Investigative Site, Piešťany, Slovak Republic
  - Novartis Investigative Site, Lučenec, Slovakia
- Thailand (4):
  - Novartis Investigative Site, Bangkok, Bangkok
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
  - Novartis Investigative Site, Khon Kaen
- United Kingdom (5):
  - Novartis Investigative Site, London, England
  - Novartis Investigative Site, Cannock, Staffordshire
  - Novartis Investigative Site, Bradford, West Yorkshire
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, London

REFERENCES:
- [Derived] Mease PJ, Kavanaugh A, Reimold A, Tahir H, Rech J, Hall S, Geusens P, Pellet P, Delicha EM, Pricop L, Mpofu S; FUTURE 1 study group. Secukinumab Provides Sustained Improvements in the Signs and Symptoms of Psoriatic Arthritis: Final 5-year Results from the Phase 3 FUTURE 1 Study. ACR Open Rheumatol. 2020 Jan;2(1):18-25. doi: 10.1002/acr2.11097. Epub 2019 Nov 14. PMID 31943974
- [Derived] Deodhar A, Gladman DD, McInnes IB, Spindeldreher S, Martin R, Pricop L, Porter B, Safi J Jr, Shete A, Bruin G. Secukinumab Immunogenicity over 52 Weeks in Patients with Psoriatic Arthritis and Ankylosing Spondylitis. J Rheumatol. 2020 Apr;47(4):539-547. doi: 10.3899/jrheum.190116. Epub 2019 Jun 15. PMID 31203228
- [Derived] Kavanaugh A, Mease PJ, Reimold AM, Tahir H, Rech J, Hall S, Geusens P, Wang Z, Pricop L, Mpofu S; FUTURE-1 Study Group. Secukinumab for Long-Term Treatment of Psoriatic Arthritis: A Two-Year Followup From a Phase III, Randomized, Double-Blind Placebo-Controlled Study. Arthritis Care Res (Hoboken). 2017 Mar;69(3):347-355. doi: 10.1002/acr.23111. PMID 27696786
- [Derived] Strand V, Mease P, Gossec L, Elkayam O, van den Bosch F, Zuazo J, Pricop L, Mpofu S; FUTURE 1 study group. Secukinumab improves patient-reported outcomes in subjects with active psoriatic arthritis: results from a randomised phase III trial (FUTURE 1). Ann Rheum Dis. 2017 Jan;76(1):203-207. doi: 10.1136/annrheumdis-2015-209055. Epub 2016 May 11. PMID 27169431
- [Derived] Mease PJ, McInnes IB, Kirkham B, Kavanaugh A, Rahman P, van der Heijde D, Landewe R, Nash P, Pricop L, Yuan J, Richards HB, Mpofu S; FUTURE 1 Study Group. Secukinumab Inhibition of Interleukin-17A in Patients with Psoriatic Arthritis. N Engl J Med. 2015 Oct;373(14):1329-39. doi: 10.1056/NEJMoa1412679. PMID 26422723

RESULTS

PARTICIPANT FLOW:
Groups:
- AIN457 (75 mg): Secukinumab (75mg)
- AIN457 (150 mg): Secukinumab (150 mg)
- Placebo Match for AIN457 ( 75 and 150 mg): Placebo match (for 75 and 150 mg)
Period: Overall Study
Arm/Group | AIN457 (75 mg) | AIN457 (150 mg) | Placebo Match for AIN457 ( 75 and 150 mg)
Started | 202 | 202 | 202
Completed | 155 | 167 | 154
Not Completed | 47 | 35 | 48
Not completed — Death | 2 | 0 | 0
Not completed — Withdrawal by Subject | 12 | 11 | 15
Not completed — Protocol Violation | 2 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 1
Not completed — Physician Decision | 7 | 5 | 2
Not completed — Lost to Follow-up | 1 | 3 | 4
Not completed — Lack of Efficacy | 14 | 10 | 15
Not completed — Adverse Event | 9 | 6 | 11

BASELINE CHARACTERISTICS:
Groups:
- Group 3: Placebo match (for 75 and 150 mg)
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Total
Number analyzed (Participants) | 202 | 202 | 202 | 606
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 180 | 180 | 192 | 552
  >=65 years | 22 | 22 | 10 | 54
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 106 | 106 | 330
  Male | 84 | 96 | 96 | 276

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients Achieving ACR20 Response Criteria on Secukinumab 75 or 150 mg vs. Placebo
Description: A patient will be considered as improved according the ACR20 criteria if she/he has at least 20 % improvement in the two following measures:Tender joint count,Swollen joint count and at least 3 of the following 5 measures: Patient's assessment of pain, Patient's global assessment disease activity,Physician's global assessment of disease activity, Health Assessment Questionnaire (HAQ©) score,Acute phase reactant (hsCRP or ESR)
Time Frame: Week 24
Population: Full analysis set
Measure: Number; unit: % participant
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 202 | 202 | 202
% participant | 50.5 | 50.0 | 17.3
Statistical Analysis 1: Comparison: Group 1 vs Group 3; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 5.53, 95% CI 2-sided [3.46 to 8.85]
Statistical Analysis 2: Comparison: Group 2 vs Group 3; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 5.39, 95% CI 2-sided [3.37 to 8.62]

2. Secondary Outcome: Percent of Subjects Achieving a PASI75 Response in the Subgroup of Subjects Who Have ≥3% Skin Involvement With Psoriasis at Baseline
Description: A 75% reduction in the Psoriasis Area and Severity Index (PASI) score (PASI 75) is the current benchmark of primary endpoints for most clinical trials with end points of psoriasis
Time Frame: Week 24
Population: Full Analysis Set
Measure: Number; unit: % participants acheiving goal
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 108 | 108 | 109
% participants acheiving goal | 64.8 | 61.1 | 8.3

3. Secondary Outcome: Percent of Subjects Achieving a PASI90 Response in the Subgroup of Subjects Who Have ≥3% Skin Involvement With Psoriasis at Baseline
Description: A 90% reduction in the Psoriasis Area and Severity Index (PASI) score (PASI 90) is above the current benchmark of primary endpoints for most clinical trials with endpoints of psoriasis
Time Frame: Week 24
Population: Full Analysis Set
Measure: Number; unit: % of participants acheiving goal
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 108 | 108 | 109
% of participants acheiving goal | 49.1 | 45.4 | 3.7

4. Secondary Outcome: Change From Baseline in DAS28-CRP for Secukinumab 75 or 150 mg
Description: DAS-CRP values range from 2.0 to 10.0 while higher values mean a higher disease activity. A DAS-CRP below the value of 2.6 is interpreted as Remission.DAS28 the DAS-CRP uses 28 different joints for its calculation: proximal interphalangeal joints (10 joints) metacarpophalangeal joints (10) wrists (2) elbows (2) shoulders (2) knees (2) With the above mentioned parameters, DAS-CRP is calculated as: <math>DAS-CRP=0.56 \times \sqrt{TEN28} + 0.28 \times \sqrt{SW28} + 0.36 \times \ln(CRP+1) + 0.014 \times SA+0.96</math> With: TEN28: number of joints with tenderness upon touching SW28: number of swollen joints CRP: C-reactive Protein SA: subjective assessment of disease activity by the patient during the preceding 7 days on a scale betweenn 0 and 100 ("0":no activity, "100": highest activity possible)
Time Frame: Week 24
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: units on scale
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 202 | 202 | 202
units on scale | -1.67 (0.085) | -1.62 (0.084) | -0.77 (0.123)

5. Secondary Outcome: Change From Baseline in SF36-PCS for Secukinumab 75 or 150 mg
Description: The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Time Frame: Week 24
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: units on scale
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 202 | 202 | 202
units on scale | 5.41 (0.524) | 5.91 (0.525) | 1.82 (0.715)

6. Secondary Outcome: Change From Baseline in HAQ-DI for Secukinumab 75 or 150 mg
Description: HAQ-DI, assesses a patient's level of functional ability and includes questions of fine movements of the upper extremity, locomotor activities of the lower extremity, and activities that involve both upper and lower extremities. There are 20 questions in eight categories of functioning which represent a comprehensive set of functional activities - dressing, rising, eating, walking, hygiene, reach, grip, and usual activities. The stem of each item asks over the past week "Are you able to …" perform a particular task. The patient's responses are made on a scale from zero (no disability) to three (completely disabled).
Time Frame: Week 24
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 202 | 202 | 202
units on a scale | -0.41 (0.036) | -0.40 (0.036) | -0.17 (0.047)

7. Secondary Outcome: Percent of Patients Achieving ACR50 Response Criteria on Secukinumab 75 or 150 mg vs. Placebo
Description: ACR50 = 50 % improvement in at least 3 of the 5 measures( Patient's assessment of pain, Patient's global assessment of disease activity, Physician's global assessment of disease activity, Health Assessment Questionnaire (HAQ©) score, C-reactive protein (CRP)/Erythrocyte Sedimentation Rate (ESR) and 50 % improvement in the swollen and tender joint count.
Time Frame: Week 24
Population: Full analysis set
Measure: Number; unit: % participant
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 202 | 202 | 202
% participant | 30.7 | 34.7 | 7.4

8. Secondary Outcome: Change From Baseline for Joint/Bone Structural Damage (Van Der Heijde Modified Total Sharp Score) for Secukinumab 75 and 150 mg (Pooled Doses)
Description: Measured are 44 joints for erosions: scored 0 to 5 in hands; 0 to 10 in feet;40 joints for joint space narrowing; summed for total score by two experienced readers scored every film blinded to patient identity, treatment, sequence of film. Lower score equals better outcome. With score of zero being normal. Joint structural damage change from baseline at Week 24 using non-parametric ANCOVA, Linear extrapolation. Estimate (for the difference in mean), SE are from a non-parametric ANCOVA model with the change from baseline van der Heijde total modified Sharp score as the dependent variable, treatment and randomization stratum (TNFa status -naive or IR ) as factors, and weight and baseline van der Heijde total modified Sharp score as covariates.
Time Frame: Week 24
Population: .Full analysis set.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 202 | 202 | 404
units on a scale | 0.02 (0.22) | 0.13 (0.20) | 0.57 (0.20)

9. Secondary Outcome: Percent of Patients With Dactylitis in the Subset of Subjects Who Have Dactylitis at Baseline
Time Frame: Week 24
Population: Full analysis set
Measure: Number; unit: % participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 104 | 104 | 116
% participants | 43.3 | 51.9 | 84.5

10. Secondary Outcome: Percent of Patients With Enthesitis in the Subset of Subjects Who Have Enthesitis at Baseline
Time Frame: Week 24
Population: Full Analysis set
Measure: Number; unit: % participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 129 | 126 | 102
% participants | 51.2 | 54.0 | 87.2

ADVERSE EVENTS:
Groups:
- Any AIN457 75 mg: Any AIN457 75 mg. After week 24 all placebo non responders were re-randomized to either 75 mg or 150 mg 1:1 to complete the trial
- Any AIN457 150 mg: Any AIN457 150 mg. After week 24 all placebo non responders were re-randomized to either 75 mg or 150 mg 1:1 to complete the trial
- Placebo: Placebo. After week 24, only reponders continued to receive placebo to the end of the trial.
Arm/Group | Any AIN457 75 mg | Any AIN457 150 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 32/292 | 51/295 | 11/202
Other Adverse Events (participants affected / at risk) | 217/292 | 222/295 | 101/202
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Any AIN457 75 mg (N=292) | Any AIN457 150 mg (N=295) | Placebo (N=202)
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 2 | 0
Angina pectoris (Cardiac disorders) | 1 | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 2 | 1
Myocardial infarction (Cardiac disorders) | 2 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 2 | 0 | 0
Goitre (Endocrine disorders) | 1 | 0 | 0
Ocular myasthenia (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Femoral hernia (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0
Impaired healing (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 2 | 1
Peripheral swelling (General disorders) | 1 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Chronic hepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | 0
Abdominal sepsis (Infections and infestations) | 1 | 0 | 0
Appendiceal abscess (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 0
Dengue fever (Infections and infestations) | 1 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 2 | 0
Erysipelas (Infections and infestations) | 1 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1 | 0
Lung abscess (Infections and infestations) | 0 | 1 | 0
Necrotising fasciitis (Infections and infestations) | 1 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 0
Prostatitis Escherichia coli (Infections and infestations) | 1 | 0 | 0
Rash pustular (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 2 | 0 | 0
Septic shock (Infections and infestations) | 2 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1
Typhoid fever (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0
Wound infection staphylococcal (Infections and infestations) | 0 | 1 | 0
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 0
Traumatic liver injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 4 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pleomorphic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Hemiplegia (Nervous system disorders) | 1 | 0 | 0
Intracranial venous sinus thrombosis (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0
Thrombotic stroke (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 2 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Any AIN457 75 mg (N=292) | Any AIN457 150 mg (N=295) | Placebo (N=202)
Anaemia (Blood and lymphatic system disorders) | 7 | 4 | 6
Leukopenia (Blood and lymphatic system disorders) | 6 | 4 | 2
Vertigo (Ear and labyrinth disorders) | 3 | 10 | 0
Dry eye (Eye disorders) | 4 | 6 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 6 | 2
Constipation (Gastrointestinal disorders) | 6 | 8 | 1
Diarrhoea (Gastrointestinal disorders) | 21 | 21 | 6
Dyspepsia (Gastrointestinal disorders) | 7 | 14 | 3
Gastritis (Gastrointestinal disorders) | 4 | 6 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 | 7 | 3
Mouth ulceration (Gastrointestinal disorders) | 5 | 9 | 0
Nausea (Gastrointestinal disorders) | 16 | 11 | 2
Toothache (Gastrointestinal disorders) | 7 | 1 | 3
Vomiting (Gastrointestinal disorders) | 12 | 4 | 1
Fatigue (General disorders) | 11 | 9 | 5
Malaise (General disorders) | 6 | 2 | 0
Oedema peripheral (General disorders) | 4 | 6 | 0
Pyrexia (General disorders) | 6 | 7 | 2
Seasonal allergy (Immune system disorders) | 5 | 6 | 0
Bronchitis (Infections and infestations) | 14 | 21 | 6
Cellulitis (Infections and infestations) | 6 | 5 | 1
Conjunctivitis (Infections and infestations) | 5 | 9 | 0
Gastroenteritis (Infections and infestations) | 8 | 20 | 2
Influenza (Infections and infestations) | 12 | 10 | 2
Lower respiratory tract infection (Infections and infestations) | 5 | 6 | 0
Nasopharyngitis (Infections and infestations) | 61 | 54 | 11
Oral herpes (Infections and infestations) | 7 | 12 | 2
Paronychia (Infections and infestations) | 4 | 8 | 0
Pharyngitis (Infections and infestations) | 10 | 14 | 0
Respiratory tract infection (Infections and infestations) | 1 | 6 | 0
Rhinitis (Infections and infestations) | 4 | 7 | 0
Sinusitis (Infections and infestations) | 10 | 16 | 4
Tinea pedis (Infections and infestations) | 6 | 2 | 0
Tonsillitis (Infections and infestations) | 8 | 2 | 0
Tooth abscess (Infections and infestations) | 8 | 8 | 0
Upper respiratory tract infection (Infections and infestations) | 52 | 60 | 12
Urinary tract infection (Infections and infestations) | 14 | 17 | 2
Viral upper respiratory tract infection (Infections and infestations) | 9 | 12 | 5
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 6 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 6 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 4 | 6 | 0
Laceration (Injury, poisoning and procedural complications) | 8 | 11 | 3
Ligament sprain (Injury, poisoning and procedural complications) | 4 | 6 | 0
Muscle strain (Injury, poisoning and procedural complications) | 6 | 8 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 3 | 8 | 1
Alanine aminotransferase increased (Investigations) | 5 | 7 | 4
Diabetes mellitus (Metabolism and nutrition disorders) | 6 | 3 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 10 | 12 | 8
Hypercholesterolaemia (Metabolism and nutrition disorders) | 11 | 15 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 | 17 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 6 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 29 | 22 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 5 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 5 | 6 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 6 | 2
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 15 | 14 | 2
Spinal pain (Musculoskeletal and connective tissue disorders) | 9 | 9 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 9 | 4 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 6 | 0
Dizziness (Nervous system disorders) | 7 | 7 | 1
Headache (Nervous system disorders) | 27 | 25 | 7
Hypoaesthesia (Nervous system disorders) | 3 | 8 | 0
Paraesthesia (Nervous system disorders) | 8 | 1 | 2
Anxiety (Psychiatric disorders) | 3 | 8 | 0
Depression (Psychiatric disorders) | 11 | 6 | 5
Insomnia (Psychiatric disorders) | 8 | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 17 | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 15 | 11 | 4
Dermatitis (Skin and subcutaneous tissue disorders) | 3 | 7 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 3 | 3
Psoriasis (Skin and subcutaneous tissue disorders) | 22 | 11 | 1
Rash (Skin and subcutaneous tissue disorders) | 8 | 8 | 7
Hypertension (Vascular disorders) | 21 | 18 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.